CLINICAL TRIAL: NCT03532672
Title: A Single Arm Trial Investigating the Acute Effect of Fasting on Metabolic, Inflammatory, and Behavioral Responses in Females With and Without Obesity
Brief Title: Early Effect of Fasting on Metabolic, Inflammatory, and Behavioral Responses in Females With and Without Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Adaliene Versiani M. Ferreira, Principal Investigator, Associate Professor, PhD, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Acute72774617.6.0000.5149
Record Dates: First submitted 2018-05-07; First posted 2018-05-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Obese
Keywords: Acute fasting; Inflammatory response; Energy Expenditure
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute fasting (Experimental): Participants will fast overnight for 10 hours (resting period), consume a santdardized breakfast, and fast during daily activities (active period) for another 10 hours.
  Interventions: Other: Acute Fasting

INTERVENTIONS:
Other: Acute Fasting — The volunteers will fast overnight (10 hours) and breakfast will be offered (bread, butter, ham and industrialized fruit juice). The participants will fast for another 10 hours during daily activities.

SUMMARY:
The aim of this study is to investigate the effect of overnight fasting versus a diurnal fasting (during daily life activities) in females with and without obesity on inflammation, neurotrophins, energy metabolism, mood, food cravings, and appetite sensations.

This study will be an acute fasting intervention.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.5 and 24.9 kg/m² or equal or greater 35 kg/m²;
* Able to sign the informed consent.

Exclusion Criteria:

* Chronic health conditions (e.g., cancer, renal, heart or liver disorders, and autoimmune diseases), or history of thyroid alterations or use of related medications;
* Use of corticosteroids, immunosuppressors, anti-inflammatories, hypoglycemics, medications for weight loss, or any medication known to interfere with metabolic and inflammatory processes (e.g., corticosteroids, nonsteroidal anti-inflammatory drugs);
* Previous surgery for weight loss;
* Inability to eat any of the components of the standardized breakfast
* Pregnancy or breastfeeding;
* Smokingç
* Alcohol use (>2 doses/day).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Blood glucose | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in blood glucose will be assessed at baseline and after 10 hours of fasting during daily activities
Lipid panel | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in lipid panel (i.e. total cholesterol, LDL, HDL and triglycerides) will be assessed at baseline and after 10 hours of fasting during daily activities
Interleukin 6 | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in blood interleukin-6 will be assessed at baseline and after 10 hours of fasting during daily activities
Appetite sensations | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in hunger, satiety, fullness, and prospective food consumption will be assessed at baseline and after 10 hours of fasting during daily activities using a 100 mm visual analogue scale
Mood states | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in anger, confusion, depression, fatigue, tension, and vigor will be assessed using the Brunel Mood Scale

SECONDARY OUTCOMES:
Gastrointestinal peptides | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in resting energy expenditure will be assessed at baseline and after 10 hours of fasting during daily activities using indirect calorimetry
Free fatty acids | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in free fatty acids will be assessed at baseline and after 10 hours of fasting during daily activities
Neurotrophic factors | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in brain-derived neurotrophic factor (BDNF), glial cell line-derived neurotrophic factor (GDNF), and nerve growth factor (NGF) will be assessed at baseline and after 10 hours of fasting during daily activities

OTHER OUTCOMES:
High-sensitivity C-reactive protein | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in blood high-sensitivity C-reactive protein will be assessed at baseline and after 10 hours of fasting during daily activities
Tumor necrosis factor-α | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in tumor necrosis factor-α will be assessed at baseline and after 10 hours of fasting during daily activities
Interleukin 8 | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in blood interleukin 8 will be assessed at baseline and after 10 hours of fasting during daily activities
Interleukin 10 | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in blood interleukin 10 will be assessed at baseline and after 10 hours of fasting during daily activities
Insulin | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in insulin will be assessed at baseline and after 10 hours of fasting during daily activities
Neutrophil/leukocyte ratio (NLR) | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in NLR will be assessed at baseline and after 10 hours of fasting during daily activities
Resting energy expenditure | At baseline (after overnight fasting) and end (after 10 hours of fasting during the day) of the intervention period (~12 hours)
  Changes in resting energy expenditure will be assessed at baseline and after 10 hours of fasting during daily activities using indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Adaliene Versiani Matos Ferreira, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Hospital das Clínicas da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tibaes JRB, Fagundes GB, Martins LB, Rodrigues AMDS, Campos AC, de Souza Cordeiro LM, Teixeira AL, Ferreira AVM. Effects of a single 10-hour daytime fasting intervention on mood and appetite in female adults with and without obesity: a real-world feasibility trial. Nutr Neurosci. 2025 Nov;28(11):1372-1385. doi: 10.1080/1028415X.2025.2514490. Epub 2025 Jun 10. PMID 40491423